CLINICAL TRIAL: NCT05110248
Title: Research and Development of Novel Quantitative Magnetic Resonance Imaging (MRI) Techniques in a Single Scan for Multiple Organ Application (RADIUS)
Brief Title: Research and Development of Novel Quantitative Magnetic Resonance Imaging (MRI) Techniques in a Single Scan for Multiple Organ Application
Acronym: RADIUS
Status: Recruiting | Type: Observational
Sponsor: Perspectum (Industry)
Responsible Party: Sponsor
Other Study IDs: 21/WS/0066
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Multiple

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cross-sectional observational study to improve MRI data acquisition techniques by optimising MRI sequences for multiple organs and assessing the repeatability and reproducibility of multiparametric MRI, in healthy volunteers.

DETAILED DESCRIPTION:
This will be a cross-sectional, observational study recruiting up to 200 healthy participants designed at improving MRI data acquisition techniques by optimising MRI sequences and assessing different aspects of the repeatability and reproducibility of multiparametric MRI. Participants will be recruited from Perspectum's own networks, as well as through advertisements on social media platforms (e.g. Facebook, Instagram), Perspectum's website, as well as through charities.

Suitable participants will be invited to attend a screening visit, normally over the telephone, which will involve collection of participant's self-reported medical evaluation to assess eligibility according to the inclusion and exclusion criteria.Visit 1 will consist of the collection of basic anthropometric measurements (e.g. height, weight, waist circumference), a medical history, and a MRI scan. Visit 2 will be a repeat of Visit 1.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Any contraindication to magnetic resonance imaging (incl. pregnancy, nonremovable electronic implants including cochlear implants, infusion pumps, and pacemakers, shrapnel injury, severe claustrophobia, allergic reaction to contrast agents)
* Any other cause, including a significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the participant's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be adult volunteers aged 18 and over, without a contraindication to magnetic resonance imaging.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Development of MRI sequences | 2 years from study start
  Development of sequences which will be used to collect good quality data on multiple organs across different MRI scanners and to ensure that desirable images are obtained within reasonable amount of time.

SECONDARY OUTCOMES:
Sequence and parameter validation | 2 years from study start
  Validation of a list of sequences and parameter details
Assessment of MRI metric repeatability | 2 years from study start
  Assessment of repeatability of the MRI metrics across 2 separate MRI acquisitions on the same scanner using statistical methods
Assessment of MRI metric reproducibility | 2 years from study start
  Assessment of reproducibility of the MRI metrics in the same participants scanned on separate MRI scanners

CONTACTS AND LOCATIONS:
Locations (1):
- Gemini One, 5520 John Smith Drive, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No